CLINICAL TRIAL: NCT00531076
Title: Phase I Study of Concurrent Bevacizumab (Avastin) With Involved-field Thoracic Radiotherapy for Inoperable Non-squamous Non-small Cell Lung Cancer, Followed by Both Concurrent and Maintenance Bevacizumab
Brief Title: Safety Study of Bevacizumab (Avastin) With Thoracic Radiation in Non-small Cell Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to toxicity
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Professor Suresh Senan, VU Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VUMC 2006/194; NL13724.029.06; EudraCTnumber 2006-003149-17
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-01

CONDITIONS: Toxicity
Keywords: bevacizumab; thoracic radiotherapy; locally-advanced non-small cell lung cancer
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: bevacizumab — Intravenous bevacizumab at 7.5mg/kg and 15mg/kg concurrently with thoracic radiotherapy in sequential cohorts.
  In the final dose level, bevacizumab 15mg/kg concurrent with radiation will be followed by maintenance bevacizumab 15mg/kg up to a maximum of 6 cycles
  Other Names: Avastin

SUMMARY:
In spite of the use of radiation combined with conventional chemotherapy, the long-term survival prognosis for most patients with locally advanced non-small cell lung cancer is disappointing. Much effort is currently focussed on exploring new molecular targeted agents that may improve upon survival. The addition of an agent that targets blood vessel formation in tumors, bevacizumab or Avastin, to conventional chemotherapy has been shown to improve survival in metastatic non-small cell lung cancer. Data from animal studies have shown that bevacizumab and related agents also increase tumor cure rates when administered both during and after radiotherapy. This suggests that combined bevacizumab and chemo-radiation may improve survival in local-advanced disease as well. Before such clinical studies can commence, the safety and normal tissue toxicity profile of bevacizumab with thoracic radiotherapy must first be established. In this study, escalating doses of bevacizumab will be administered during radiotherapy, followed by maintenance bevacizumab.

ELIGIBILITY:
Inclusion criteria:

1. Cytologically or histologically confirmed stages II or III non-squamous NSCLC
2. No evidence of tumour invading major blood vessels and no active hemoptysis (bright red blood of at least ½ teaspoon) in the 28 days prior to randomization.
3. No prior systemic therapy for NSCLC. Prior surgery and/or extra-thoracic irradiation is permitted.
4. Presence of at least one measurable target lesion
5. Age 18 or greater.
6. WHO performance status of 0 or 1.
7. Acceptable pulmonary function as defined by a Fev1 of ≥30% and a DLCO of ≥40% of predicted
8. Life expectancy of at least 12 weeks.
9. Adequate hematological, renal and hepatic functions

   * Absolute neutrophil count >2x109/l.
   * Platelet count > 100x109/l.
   * Total bilirubin < 1.5 x UNL
   * ASAT/ALAT < 2 x UNL
   * Alkaline phosphatase < 5 x UNL
   * Creatinine < 130 μmol/L
   * Creatinine clearance > 60 ml/min; measured or calculated
10. Urine dipstick for proteinuria < 1+. If urine dipstick is ≥ 1, 24 hour urine must demonstrate < 500 mg of protein in 24 hours.
11. No pre-existing sensory neurotoxicity grade 2 (CTC)
12. No active (uncontrolled) infection requiring antibiotics

Exclusion criteria:

1. Mixed tumor types with small cell lung cancer or squamous cell carcinoma
2. Other serious diseases, such as heart failure, angina pectoris, myocardial infarction within the last 6 months, uncontrolled hypertension
3. Serious non-healing wound or ulcer.
4. ASAT and ALAT > 1,5 x UNL
5. alkaline phosphatase 5 x UNL
6. Evidence of bleeding diathesis or coagulopathy.
7. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed with the patient before registration in the trial.
8. Participation in other trial with investigational drug or treatment modality.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To establish the safety and tolerability of 2 dose-levels of bevacizumab administered every 3 weeks with concurrent thoracic radiotherapy to 66 Gy,and also maintenance (15 mg/kg) bevacizumab following completion of thoracic radiotherapy | 1 year

SECONDARY OUTCOMES:
Correlate all observed toxicity with dose-volume histograms of irradiated normal organs and explore surrogate tumor end-points that may correlate with the efficacy of combined treatment with anti-VEGF targeted therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Suresh Senan, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Egbert F Smit, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands